CLINICAL TRIAL: NCT07352319
Title: Effects of Lower Body Plyometric Training on Serum CPK and Creatinine Levels in Collegiate Female Volleyball Players: An Experimental Study
Brief Title: DOES LOWER BODY PLYOMETRICS CAUSE RHABDOMYOLYSIS IN FEMALE VOLLEYBALL PLAYERS-AN EXPERIMENTAL STUDY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Elsayed Mohamed Abd Alaal, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BMC VP
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Exercise-Induced Muscle Damage; Rhabdomyolysis; Athletes
MeSH Terms: conditions — Rhabdomyolysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lower-body plyometric training (Experimental): Progressive plyometric program, twice weekly for eight weeks.
  Interventions: Other: plyometric program
- Control (Active Comparator): Routine volleyball practice; no plyometric exercises.
  Interventions: Other: plyometric program

INTERVENTIONS:
Other: plyometric program — Twice-weekly sessions (Mon/Wed) for 8 weeks; exercise menu and dosing per Table 1 (intensity, rest, and jumps/set).
  Other Names: Lower-body plyometric training

SUMMARY:
Eight-week interventional study to evaluate whether lower-body plyometric training alters serum creatine phosphokinase (CPK) and creatinine levels in female collegiate volleyball players. Sixty participants were randomized to experimental (plyometrics twice weekly) or control (routine volleyball) groups. Blood sampling occurred at baseline; days 2, 4, and 6; and weeks 1, 2, 4, 6, and 8.

DETAILED DESCRIPTION:
Intervention adapted from James & Robert (2015). Experimental group completed progressive lower-body plyometrics twice weekly (Monday/Wednesday) over eight weeks with warm-up and cool-down. Exercises included squat jump; jump to box (30 cm); tuck jump; split squat jump; lateral hurdle jump (50 cm); zigzag jump; single-leg tuck jump; and depth jump (80 cm). Control group continued routine volleyball activities and did not perform low/medium/high-intensity plyometrics. Primary biomarker (serum CPK) assessed via CK-NAC optimized IFCC method; serum creatinine by modified Jaffe's method. Two-way ANOVA with Bonferroni post hoc used. Findings: CPK increased from day 2, peaked day 4, stabilized to week 2, then declined toward baseline by week 8; creatinine remained stable.

ELIGIBILITY:
Inclusion Criteria:

Active collegiate female volleyball players

* consent to participate
* no prior plyometric training program.

Exclusion Criteria:

* Neuromuscular impairments
* recent injuries.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Serum CPK (U/L) | Baseline; 2, 4, 6 days; 1, 2, 4, 6, 8 weeks
  change from baseline at day 2, day 4, week 1, week 2, week 4, week 6, week 8

SECONDARY OUTCOMES:
Serum creatinine (mg/dL) | Baseline; 2, 4, 6 days; 1, 2, 4, 6, 8 weeks
  change from baseline over same time points

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Mariam Salem, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because this study does not include a data-sharing plan and is limited to internal analysis only.